CLINICAL TRIAL: NCT06628960
Title: The Effect of Su Jok Therapy on Breastfeeding Success, Breastfeeding Self-Efficacy and Perception of Insufficient Milk After Caesarean Section in Primiparas
Brief Title: Effect of Su Jok Therapy on Breastfeeding
Acronym: Sujok
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aysegul Kilicli (Other)
Responsible Party: Sponsor-Investigator, Aysegul Kilicli, Gaziantep University, University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MAUN
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Breastfeeding
Keywords: Su Jok therapy; cesarean section; breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- su jok therapy; (Experimental): su jok therapy; application of seeds placed at certain points on the palm of the hand every day for the first ten days after birth, every day to be kept in the hand for 2 hours.
  Interventions: Behavioral: Su Jok Therapy
- control group (No Intervention): control group, Su Jok will not be applied

INTERVENTIONS:
Behavioral: Su Jok Therapy — Su Jok Therapy
  Arms: su jok therapy;

SUMMARY:
There are many alternative methods to increase breast milk. In the literature, studies on Su Jok therapy applications are limited and no studies on increasing breast milk have been found. In Korean language, 'Su' means hand and 'Jok' means foot. Su Jok therapy is defined as a modern acupressure/acupuncture interpretation that utilises the body's independent communication systems on the hands and feet by applying various techniques such as massage, moxa (heating), needles, magnets and seeds to the reflection points on the hands and feet. Su Jok is an integrated therapy that incorporates many tried and trusted methods of oriental medicine

DETAILED DESCRIPTION:
There are many alternative methods to increase breast milk. In the literature, studies on Su Jok therapy applications are limited and no studies on increasing breast milk have been found. In Korean language, 'Su' means hand and 'Jok' means foot. Su Jok therapy is defined as a modern acupressure/acupuncture interpretation that utilises the body's independent communication systems on the hands and feet by applying various techniques such as massage, moxa (heating), needles, magnets and seeds to the reflection points on the hands and feet. Su Jok is an integrated therapy that incorporates many tried and trusted methods of oriental medicine.

ELIGIBILITY:
Inclusion Criteria:

* primiparous women giving birth by caesarean section,
* women aged 19-35,
* breastfeeding women

Exclusion Criteria:

* those who refused to participate in the research

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — primiparous women giving birth by caesarean section, women aged 19-35, breastfeeding women
Enrollment: 60 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy Scale | pre-test
  It was developed by Dennis (2003). Its Turkish validity and reliability was conducted by Aluş Tokat et al. (2010). The scale consists of 14 items and is in five-point Likert type. A minimum of 14 points and a maximum of 70 points can be obtained from the scale. All items are positive. A minimum of 14 points and a maximum of 70 points can be obtained from the scale. All items are positive. The higher the score obtained from the scale, the higher the breastfeeding self-efficacy.
Breastfeeding Self-Efficacy Scale | 3rd day after caesarean section
  It was developed by Dennis (2003). Its Turkish validity and reliability was conducted by Aluş Tokat et al. (2010). The scale consists of 14 items and is in five-point Likert type. A minimum of 14 points and a maximum of 70 points can be obtained from the scale. All items are positive. A minimum of 14 points and a maximum of 70 points can be obtained from the scale. All items are positive. The higher the score obtained from the scale, the higher the breastfeeding self-efficacy.
Breastfeeding Self-Efficacy Scale | 10th day after caesarean section
  It was developed by Dennis (2003). Its Turkish validity and reliability was conducted by Aluş Tokat et al. (2010). The scale consists of 14 items and is in five-point Likert type. A minimum of 14 points and a maximum of 70 points can be obtained from the scale. All items are positive. A minimum of 14 points and a maximum of 70 points can be obtained from the scale. All items are positive. The higher the score obtained from the scale, the higher the breastfeeding self-efficacy.
Breastfeeding Charting System: LATCH | pre-test
  It was developed by Jensen et al. (1994). Its Turkish validity and reliability was performed by Yenal and Okumuş (2003). LATCH includes five evaluation criteria and consists of the first letters of the English equivalents of these criteria. In the LATCH Scoring System, 0, 1 or 2 points are given for each criterion A minimum score of 0 and a maximum score of 10 can be obtained from the scale. All items are positive. The higher the score obtained from the scale, the higher the breastfeeding self-efficacy.
Breastfeeding Charting System: LATCH | 3rd day after caesarean section
  It was developed by Jensen et al. (1994). Its Turkish validity and reliability was performed by Yenal and Okumuş (2003). LATCH includes five evaluation criteria and consists of the first letters of the English equivalents of these criteria. In the LATCH Scoring System, 0, 1 or 2 points are given for each criterion. A minimum score of 0 and a maximum score of 10 can be obtained from the scale. All items are positive. The higher the score obtained from the scale, the higher the breastfeeding self-efficacy.
Breastfeeding Charting System: LATCH | 10th day after caesarean section
  It was developed by Jensen et al. (1994). Its Turkish validity and reliability was performed by Yenal and Okumuş (2003). LATCH includes five evaluation criteria and consists of the first letters of the English equivalents of these criteria. In the LATCH Scoring System, 0, 1 or 2 points are given for each criterion. A minimum score of 0 and a maximum score of 10 can be obtained from the scale. All items are positive. The higher the score obtained from the scale, the higher the breastfeeding self-efficacy.
Inadequate Milk Perception Scale | pre-test
  The scale developed by McCarter-Spaulding and Kearney in 2001 consists of 6 questions to determine inadequate perception of breast milk. The first question questioning whether the mother perceives her milk as sufficient or not is in the form of 'yes' or 'no'. The other 5 questions aim to measure the perception of inadequacy of milk and are scored between 0-10. '0' indicates that milk is perceived as completely inadequate and "10" indicates that milk is perceived as completely adequate. The scale is scored between 0-50. A high score indicates an increased perception of milk sufficiency.
Inadequate Milk Perception Scale | 3rd day after caesarean section
  The scale developed by McCarter-Spaulding and Kearney in 2001 consists of 6 questions to determine inadequate perception of breast milk. The first question questioning whether the mother perceives her milk as sufficient or not is in the form of 'yes' or 'no'. The other 5 questions aim to measure the perception of inadequacy of milk and are scored between 0-10. '0' indicates that milk is perceived as completely inadequate and "10" indicates that milk is perceived as completely adequate. The scale is scored between 0-50. A high score indicates an increased perception of milk sufficiency.
Inadequate Milk Perception Scale | 10th day after caesarean section
  The scale developed by McCarter-Spaulding and Kearney in 2001 consists of 6 questions to determine inadequate perception of breast milk. The first question questioning whether the mother perceives her milk as sufficient or not is in the form of 'yes' or 'no'. The other 5 questions aim to measure the perception of inadequacy of milk and are scored between 0-10. '0' indicates that milk is perceived as completely inadequate and "10" indicates that milk is perceived as completely adequate. The scale is scored between 0-50. A high score indicates an increased perception of milk sufficiency.

CONTACTS AND LOCATIONS:
Overall Officials: AYŞEGÜL KILIÇLI, Assisstan. Prof. PhD., Principal Investigator — Muş Alparslan University
Locations (1):
- Şanlıurfa training and research hospital, Sanliurfa, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 15 October 2024- 15 October 2025
Access Criteria: 15 October 2024- 15 October 2025